CLINICAL TRIAL: NCT06965790
Title: Randomized Controlled Study on Sex-specific, Individualized Dose Calculation of Intravenously Administered Contrast Agent in CT Examinations in Portal Venous Phase to Achieve Equivalent Contrast in Men and Women
Brief Title: Study on Sex-specific, Individualized Dose Calculation of Contrast Agent in CT Examinations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24040
Record Dates: First submitted 2025-03-25; First posted 2025-05-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: CT Scans; Contrast Media; Gender; Womens Health
Keywords: CT; CT Scans; Contrast Media; contrast; gender
MeSH Terms: conditions — Coitus | interventions — Contrast Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight adjusted contrast media volume (No Intervention): control group with regular weight adjusted dosing
- blood volume adjusted contrast media volume (Active Comparator): study group with dosing according to sex-specific blood volume
  Interventions: Drug: contrast media (Imeron 350, active ingredient Iomeprol) volume according to sex-specific blood volume

INTERVENTIONS:
Drug: contrast media (Imeron 350, active ingredient Iomeprol) volume according to sex-specific blood volume — Calculation of the standardized contrast agent (Imeron 350, active ingredient Iomeprol) quantity (0.35 g iodine/kg) and calculation of the specific blood volume using the established Nadler formula for male and female. Adjustment of the contrast agent according to the ratio of the blood volumes. The amount of saved contrast agent is replaced 1:1 by NaCl.
  Arms: blood volume adjusted contrast media volume

SUMMARY:
A large proportion of radiological CT examinations require the intravenous administration of iodine-containing X-ray contrast medium. According to current guidelines, the amount required for CT examinations in the (portal) venous phase is calculated on the basis of body weight (e.g. 0.2-0.4 g iodine/kg body weight), but a standardized application dose of the contrast agent is often also used.

In earlier studies, the investigators found that the iodine contrast in vessels and organs achieved with a standardized amount of contrast agent differs significantly between women and men. On average, women showed around 10% higher iodine contrast than men of the same height and weight. The investigators attribute these differences to physiological, sex-specific differences in blood volume. For example, the blood volume of a woman 175 cm tall and weighing 75 kg is approx. 400 ml less than that of a man of the same height and weight (approx. 4.6 vs. 5.0 l, calculated according to Nadler). Taking blood volume into account, sex was no longer a significant influencing factor in a retrospective cohort (n=274).

The investigators would now like to investigate these results in a prospective study. For this purpose, two groups of patients with a clinical indication for a contrast-enhanced CT scan in the venous phase will be compared:

1. control group with regular weight-adjusted (n = 200)
2. study group with dosing according to blood volume (n = 200).

The hypothesis is that the application scheme adapted to the blood volume leads to a more homogeneous contrasting of women and men. In order to quantify this effect, the iodine contrast values of both groups will be quantitatively analyzed, taking into account other influencing variables (height, weight).

The investigators hope that this approach will reduce or even eliminate the observed sex-specific differences. This would lead to a sex-equal contrast based on an individualized amount of contrast medium.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a justifying indication for a CT scan of the thorax and abdomen with application of intravenous contrast medium and a start delay corresponding to the portal venous contrast medium phase
* Ability to give informed consent, as well as written and verbal consent to participate in the study available

Exclusion Criteria:

* Cardiorespiratory instability (as assessed by the attending physician)
* Age <18 years
* Existing or suspected pregnancy
* Known post hepatectomy and/or splenectomy
* Lack of current height (in the same inpatient/outpatient hospital stay) or lack of possibility of height measurement
* Lack of current daily body weight or inability to measure body weight
* Height under 140 cm or over 220 cm
* Body weight under 50 kg or over 120 kg
* Contraindication to iodine-containing contrast medium (Allergy to contrast media containing iodine, Severe renal insufficiency (eGFR < 30 ml/min), Hyperthyroidism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sex-specific contrast difference in the vessels and organs | 1 year
  Achieved iodine contrast (Hounsfield units) in vessels and organs
Contrasting the organs after adjusting the application dose of the contrast agent to the specific blood volume | 1 year
  Achieved iodine contrast (Hounsfield units) in vessels and organs

SECONDARY OUTCOMES:
Evaluation of whether the adapted blood volume formula according to Nadler can be used to achieve the minimum amount of contrast medium required to ensure sufficient contrast | 1 year
  Quantitative measurements of the attenuation of the liver, the portal vein, the aorta, the spleen and the kidneys by placing circular ROIs on CT-series. Mean and standard deviation of CT-values are obtained from contrast enhanced series, iodine maps and virtual non-contrast series. The measurements are performed by blinded physicians using anonymized data on a dedicated workstation.
Evaluation of the contrast values achieved that still allow sufficient assessment of the vessels and organs. | 1 year
  Quantitative measurements of the attenuation of the liver, the portal vein, the aorta, the spleen and the kidneys by placing circular ROIs on CT-series. Mean and standard deviation of CT-values are obtained from contrast enhanced series, iodine maps and virtual non-contrast series. The measurements are performed by blinded physicians using anonymized data on a dedicated workstation.
Comparison of the diagnostic accuracy of DECT/MECT-based imaging of vascular and organ structures. | 1 year
  Quantitative measurements of the attenuation of the liver, the portal vein, the aorta, the spleen and the kidneys by placing circular ROIs on CT-series. Mean and standard deviation of CT-values are obtained from contrast enhanced series, iodine maps and virtual non-contrast series. The measurements are performed by blinded physicians using anonymized data on a dedicated workstation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hosptial Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No